CLINICAL TRIAL: NCT03803566
Title: Age-independent Decline in Manual Dexterity of Middle-aged and Older Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The grant application has not been approved
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Roger Enoka, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-0269
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Aging
Keywords: Manual dexterity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faster (Experimental): This group will comprise participants who complete the grooved pegboard test at baseline with a time of less than 71 seconds. One half of the members in this group will perform the two interventions in the order of pegboard practice and then force control practice, whereas the other half of the group will perform the two practice interventions in the opposite order.
  Interventions: Other: Pegboard practice; Other: Force control practice
- Slower (Experimental): This group will comprise participants who complete the grooved pegboard test at baseline with a time of greater than 70 seconds. One half of the members in this group will perform the two interventions in the order of pegboard practice and then force control practice, whereas the other half of the group will perform the two practice interventions in the opposite order.
  Interventions: Other: Pegboard practice; Other: Force control practice

INTERVENTIONS:
Other: Pegboard practice — Practice of the grooved pegboard test
Other: Force control practice — Practice performing steady muscle contractions

SUMMARY:
The objective of the clinical trial is to evaluate the mediating influence of force control on the pegboard times of adults (50-89 years) who are stratified into groups of faster and slower pegboard times. The hypothesis is that practice of either a pegboard test or a force-control task will reduce pegboard times, but the decrease will be greater and less similar after the two practice interventions for the slower group of participants. The outcomes are expected to demonstrate that force control is a modifiable mediator of pegboard times for this cohort, but the effect will be stronger for the group with faster pegboard times.

DETAILED DESCRIPTION:
The study will involve a randomized, cross-over design with a one-week washout between arms. The two arms (3 weeks each) will comprise practice of the grooved pegboard test and practice of steady contractions while lifting and lowering light loads with a hand muscle. Randomization into practice order will be accomplished with a block approach (block size = 4) for each of the two groups. The outcome assessors will be blinded to practice order. The outcomes will comprise three tests of manual dexterity and the measurement of force control during submaximal contractions. The outcomes will be obtained before and after the six sessions in each practice arm.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, and speak English
* Able to arrange transportation to the Boulder campus

Exclusion Criteria:

* Cognitive impairment
* Major psychiatric condition
* Unstable depressive disorder
* Progressive neurological, muscular, cardiovascular, or skeletal disorder
* Chronic pain condition
* Currently taking medication known to influence neuromuscular function
* Recent hospitalization
* Unable to attend 12 practice sessions in 6 weeks

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Grooved pegboard test | Changes from baseline (week 1) at weeks 4 and 7
  Time to complete the test as quickly as possible
9-hole pegboard test | Changes from baseline (week 1) at weeks 4 and 7
  Time to complete the test as quickly as possible
Jebsen Hand Function test | Changes from baseline (week 1) at weeks 4 and 7
  Time to complete the test as quickly as possible
Force control | Changes from baseline (week 1) at weeks 4 and 7
  The coefficient of variation for force when subjects exert a constant submaximal force

SECONDARY OUTCOMES:
EMG amplitude | Changes from baseline (week 1) at weeks 4 and 7
  Absolute amplitude of the electromyographic (EMG) signal for the involved muscles during the steady contractions
MVC force | Changes from baseline (week 1) at weeks 4 and 7
  The peak force exerted during a maximal isometric contractions
1-RM load | Changes from baseline (week 1) at weeks 4 and 7
  The maximal weight that can be lifted once
Index finger acceleration | Changes from baseline (week 1) at weeks 4 and 7
  The average standard deviation of index finger acceleration in the abduction-adduction plane when a light load is being lifted and lowered during the practice intervention
Motor unit discharge rates | Changes from baseline (week 1) at weeks 4 and 7
  The discharge times of action potentials by motor units during the steady submaximal contractions

CONTACTS AND LOCATIONS:
Overall Officials: Roger Enoka, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No